CLINICAL TRIAL: NCT05031975
Title: Temozolomide and Irinotecan Consolidation in Patients With MGMT Silenced, Microsatellite Stable Colorectal Cancer With Persistence of Minimal Residual Disease in Liquid Biopsy After Standard Adjuvant Chemotherapy: the ERASE-TMZ Study
Brief Title: Temozolomide and Irinotecan in Patients With MGMT Silenced Colorectal Cancer After Adjuvant Chemotherapy
Acronym: ERASE-TMZ
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 03/21
Record Dates: First submitted 2021-08-24; First posted 2021-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Colorectal Cancer
Keywords: Temozolomide; MGMT; microsatellite stable; ctDNA; TEMIRI; Stage II; Stage III; post-adjuvant
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEMIRI (Experimental): Irinotecan intravenous infusion (IV) given every 14 days in combination with oral (PO) temozolomide over days 1-5 every 28 days.
  The treatment will consist of six 28-days cycles of TEMIRI.
  Interventions: Drug: Irinotecan; Drug: Temozolomide

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 100 mg/smq intravenous infusion every 14 days
Drug: Temozolomide — Oral temozolomide 150 mg/sqm over days 1-5 every 28 days.

SUMMARY:
Surgical resection is curative for 75% of stage II and 50% of stage III colon cancer patients. The magnitude of benefit of adjuvant chemotherapy in terms of disease-free (DFS) and overall survival (OS) varies according to TNM stage and microsatellite status. Standard adjuvant chemotherapy includes fluoropyrimidine and oxaliplatin regimens for up to six months.

Circulating tumor DNA (ctDNA) detected after surgical resection reflects the presence of micrometastatic disease and pivotal observational studies addressed the prognostic value of ctDNA in the post-surgical setting. Adjuvant chemotherapy can promote the clearance of ctDNA, and ctDNA clearance after adjuvant chemotherapy is prognostic for better DFS in patients with stage III resected cancers and post-operative positive ctDNA.

ctDNA may be investigated as a potential real-time surrogate biomarker of the efficacy of adjuvant therapy, but suggest that patients with ctDNA persistence after standard chemotherapy might be "molecularly metastatic" and may benefit from additional "consolidation" non-cross resistant strategies aimed at clearing micrometastatic disease.

Temozolomide has modest but non-negligible activity (about 10%) in chemo-refractory patients with MGMT methylated mCRC. The response rate to temozolomide-based therapy in pretreated patients is increased to up to 20% when restricting the focus on those with MGMT IHC-negative/MGMT methylated and MSS cancers Significant activity (ORR 26%) and favorable safety profile were reported by the combination of temozolomide and irinotecan (TEMIRI regimen) in patients with pretreated MGMT methylated/MSS mCRC, thus suggesting that the two agents may have synergist activity in line with preclinical data.

Based on all these considerations, there is a strong rationale for investigating TEMIRI regimen as consolidation non-cross resistant therapy in a liquid-biopsy driven interventional trial.

Eligible patients with MGMT-silenced, MSS, radically resected CRC and detectable ctDNA after standard chemotherapy will be enrolled and will receive 6-month post-adjuvant/consolidation TEMIRI (given for up to 6 monthly cycles).

DETAILED DESCRIPTION:
Surgical resection is curative for 75% of stage II and 50% of stage III colon cancer patients. The magnitude of benefit of adjuvant chemotherapy in terms of disease-free (DFS) and overall survival (OS) varies according to TNM stage and microsatellite status. Specifically, in patients with stage II microsatellite stable (MSS) tumors and high risk clinical features (i.e. pT4, lymphovascular invasion, perineural invasion, bowel obstruction, positive surgical margins and inadequately sampled lymph nodes) adjuvant therapy with fluoropyrimidines conditioned a modest but significant DFS benefit, while oxaliplatin-based therapy may be offered to patients with poor prognosis such as those with pT4 disease. In patients with stage III disease adjuvant therapy with oxaliplatin and fluoropyrimidine combinations significantly improved DFS and OS in phase 3 randomized trials. However, oxaliplatin is burdened by dose-cumulative and potentially long-lasting neurotoxicity. Therefore, three-month duration of oxaliplatin-based chemotherapy was compared to six-month in six randomized trials including patients with resected stage (II)/III colon cancer. In the pooled analysis of such trials (IDEA Collaboration), the non-inferiority for DFS of three months adjuvant oxaliplatin-based chemotherapy was not formally demonstrated. However, absolute DFS loss with 3- month therapy was clearly unsignificant from a clinical point-of-view and 3-month duration of oxaliplatin-based adjuvant chemotherapy is now recommended in patients with low risk disease (pT3N1) and particularly when adopting a capecitabine-based regimen (CAPOX).

Circulating tumor DNA (ctDNA) detected after surgical resection reflects the presence of micrometastatic disease and pivotal observational studies addressed the prognostic value of ctDNA in the post-surgical setting. Detectable ctDNA after surgery is prognostic for DFS in patients with resected colon cancer with high specificity in predicting recurrence (-100%), reinforcing its promising role for guiding trials on post-surgical intensification strategies, but ctDNA is also endowed with suboptimal sensitivity (70%), thus limiting its potential usefulness to guide the complete omission of adjuvant chemotherapy. Regarding the impact of adjuvant chemotherapy on micrometastatic disease, adjuvant chemotherapy was able to clear ctDNA in individual patients with resected stage II tumors. Moreover, ctDNA clearance after adjuvant chemotherapy was prognostic for better DFS in patients with stage III resected cancers and post-operative positive ctDNA. Collectively, these data highlight that ctDNA may be investigated as a potential real-time surrogate biomarker of the efficacy of adjuvant therapy, but suggest that patients with ctDNA persistence after standard chemotherapy might be "molecularly metastatic" and may benefit from additional "consolidation" non-cross resistant strategies aimed at clearing micrometastatic disease.

Temozolomide displayed limited activity (overall response rate [ORR] 9%) in patients with heavily pretreated metastatic colorectal cancer (mCRC) with MGMT promoter methylation assessed by means of a qualitative assay - methylation-specific PCR. However, even if MGMT promoter methylation is found in up to 40% of patients with colorectal cancer, in-silico analyses and translational analyses showed that only a subset of these tumors (- 10% of all comers) display lack of MGMT expression and negative MGMT IHC staining. In keeping with findings, correlative studies of phase 2 trials showed that MGMT immunohistochemical negativity and higher MGMT methylation % by quantitative assays are associated with temozolomide activity. Finally, proficiency of the mismatch repair is needed for alkylators activity. Therefore, temozolomide might be considered a tailored chemotherapy in patients with MGMT silenced tumors (i.e. those with MGMT negative expression and MGMT promoter methylation) and microsatellite stable (MSS) tumors. Significant activity (ORR 26%) and favorable safety profile were reported by the combination of temozolomide and irinotecan (TEMIRI regimen) in patients with pretreated MGMT methylated/MSS mCRC, thus suggesting that the two agents may have synergist activity in line with preclinical data.

Moving from this rationale we designed a phase 2 proof-of-concept trial aimed at evaluating the activity in terms of ctDNA clearance or "seroreversion" after TEMIRI regimen as a post-adjuvant strategy in patients with MGMT silenced, MSS colorectal cancer (CRC) with positive ctDNA after oxaliplatin-based adjuvant standard chemotherapy.

Eligible patients with MGMT-silenced, MSS, radically resected CRC and detectable ctDNA after standard chemotherapy will be enrolled and will receive 6-month post-adjuvant/consolidation TEMIRI (given for up to 6 monthly cycles).

ELIGIBILITY:
Inclusion Criteria:

* Have provided written informed consent prior to any study specific procedures.
* Age ≥ 18 years.
* Histologically confirmed diagnosis of stage III or T4N0 stage II colon cancer (located 12 cm from the anal verge by endoscopy and above the peritoneal reflection at surgery) or histologically confirmed diagnosis of locally-advanced resectable rectal cancer (proximal margin located at < 12 cm from the anal verge).
* Radical surgery for patients with colon cancer or preoperative (chemo)-radiotherapy followed by radical surgery for patients with rectal cancer.
* Completion of at least 3 months of oxaliplatin-based (CAPOX or FOLFOX) adjuvant chemotherapy (or candidate to oxaliplatin-based adjuvant chemotherapy if post-surgery pre-screening).
* Availability of the archival FFPE tumor tissue obtained prior to any treatment.
* Acceptance to undergo all the interventional and exploratory liquid biopsies.
* Absent MGMT expression by IHC, MGMT promoter methylation by pyrosequencing (> 5%) and MSS by standard assessment.
* Presence of ctDNA in the liquid biopsies collected at 2-6 weeks after the last dose of standard adjuvant chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Completion of adjuvant chemotherapy for a duration of at least three months.
* Adequate organ function as defined below:
* Hematological function indicated by all of the following:

White Blood Cell (WBC) count ≥ 2 x 109/L Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L Hemoglobin ≥ 9 g/dL (patients may have transfusions and/or growth factors to attain adequate Hb).

- Liver function indicated by all of the following: Total bilirubin < 1.5 x upper limit of normal (ULN) Aspartate transaminase (AST) and alanine aminotransferase (ALT) < 3 x ULN Alkaline phosphatase (ALP) < 2 x ULN.

- Renal function indicated by all of the following: Serum creatinine < 1.5 x ULN or calculated creatinine clearance > 40 ml/min.

- Coagulation indicated by all of the following: INR ≤ 1.5 and aPTT ≤ 1.5 x ULN within 7 days prior to the start of study treatment for patients not receiving anti-coagulation. a. NOTE: The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least two weeks prior to the start of study treatment.

* Carcinoembryonic antigen (CEA) level ≤ 10 ng/ml.
* No evidence of distant metastases or loco-regional disease by computed tomography scan or magnetic resonance imaging.
* Male subjects with female partners of childbearing potential must be willing to use adequate contraception as approved by the investigator (barrier contraceptive measure or oral contraception).
* Women of childbearing potential must have a negative blood pregnancy test at the baseline visit and must be willing to use adequate contraception as approved by the investigator (barrier contraceptive measure or oral contraception). For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 months, are surgically sterile, or are sexually inactive.

Exclusion Criteria:

* History of another neoplastic disease, unless in remission for ≥ 5 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Had an incomplete diagnostic colonoscopy and/or polyps removal.
* Microscopic or macroscopic evidence of residual tumor (R1 or R2 resections). Patients should never have had any evidence of metastatic disease (including presence of tumor cells in the peritoneal lavage).
* Current or recent treatment with another investigational drug or participation in another investigational study.
* Inability to swallow pills.
* Active infection requiring intravenous antibiotics at the start of study treatment.
* Evidence of any other disease, neurologic or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of any of the study medications, puts the patient at higher risk for treatment-related complications or may affect the interpretation of study results.

Patient unable to comply with the study protocol owing to psychological, social or geographical reasons.

* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Sexually active males and females (of childbearing potential) unwilling to practice contraception (barrier contraceptive measure or oral contraception) during the study and until 6 months after the last trial treatment.
* Clinically significant (i.e. active) cardiovascular disease, for example cerebrovascular accidents ≤ 6 months prior to start of study treatment, myocardial infarction ≤ 6 months prior to study enrolment, unstable angina, New York Heart Association (NYHA) Functional Classification Grade II or greater congestive heart failure, or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment.
* Known presence of one of the following UGT1A1 1(TA)6/UGT1A1 36(TA)5; UGT1A1 28(TA)7/UGT1A1 37(TA)8 (homozygous genotype).
* Known presence of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
To assess the activity in terms of seroreversion of TEMIRI consolidation regimen administered to patients with high-risk stage II (pT4) or III MSS, MGMT silenced CRC and positive post-adjuvant ctDNA after standard oxaliplatin-based adjuvant chemotherapy. | 2 years from randomization
  The activity of TEMIRI will be measured as the rate of patients with post-treatment seroreversion and disease-free at 2 years

SECONDARY OUTCOMES:
Disease-free survival (DFS) of patients treated with TEMIRI as consolidation regimen | 36 months
  DFS is defined as the time from randomization to recurrence of tumor or death due to any cause, whichever occurs first. DFS will be censored on the date of the last evaluable on study tumour assessment documenting absence of disease relapse for patients who are alive and disease-free at the time of the analysis. Alive patients having no tumour assessments after baseline will have time to event censored on the data of enrolment
Overall survival (OS) of patients treated with TEMIRI as consolidation regimen | 36 months
  OS is defined as the time from enrolment to the date of death due to any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.
Safety profile of TEMIRI consolidation regimen | 36 months
  Safety will be assessed by monitoring the frequency of adverse events
Quality of life as assessed using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Assessed up to 24 months from enrollment
  EORTC QLQ-C30 administered every 12 weeks during treatment and at the date of first documented progression, assessed up to 24 months from enrollment
Quality of life as assessed using the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Colorectal Cancer 29 (EORTC QLQ-CR29) | Assessed up to 24 months from enrollment
  EORTC QLQ-CR29 administered every 12 weeks during treatment and at the date of first documented progression, assessed up to 24 months from enrollment
Quality of life as assessed using the Euro Quality of Life 5 Dimensions Questionnaire (EQ-5D-5L) | Assessed up to 24 months from enrollment
  EQ-5D-5L administered every 12 weeks during treatment and at the date of first documented progression, assessed up to 24 months from enrollment

OTHER OUTCOMES:
Identify a gene expression signature (name of mutated gene/genes) associated to temozolomide resistance/sensitivity | 36 months
  To develop a gene expression signature (a single or combined group of genes) associated with temozolomide resistance/sensitivity by profiling tumor tissue blocks obtained prior to any treatment
To assess the accuracy of ctDNA as disease recurrence biomarker | 36 months
  To longitudinally monitor the disease recurrence thanks to serial liquid biopsies obtained during the follow-up phase. The outcome will be measured as the percentage of ctDNA negative patients with recurrence disease

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Pietrantonio, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI, Italy

REFERENCES:
- [Background] Ribic CM, Sargent DJ, Moore MJ, Thibodeau SN, French AJ, Goldberg RM, Hamilton SR, Laurent-Puig P, Gryfe R, Shepherd LE, Tu D, Redston M, Gallinger S. Tumor microsatellite-instability status as a predictor of benefit from fluorouracil-based adjuvant chemotherapy for colon cancer. N Engl J Med. 2003 Jul 17;349(3):247-57. doi: 10.1056/NEJMoa022289. PMID 12867608
- [Background] Quasar Collaborative Group; Gray R, Barnwell J, McConkey C, Hills RK, Williams NS, Kerr DJ. Adjuvant chemotherapy versus observation in patients with colorectal cancer: a randomised study. Lancet. 2007 Dec 15;370(9604):2020-9. doi: 10.1016/S0140-6736(07)61866-2. PMID 18083404
- [Background] Bockelman C, Engelmann BE, Kaprio T, Hansen TF, Glimelius B. Risk of recurrence in patients with colon cancer stage II and III: a systematic review and meta-analysis of recent literature. Acta Oncol. 2015 Jan;54(1):5-16. doi: 10.3109/0284186X.2014.975839. Epub 2014 Nov 28. PMID 25430983
- [Background] Andre T, de Gramont A, Vernerey D, Chibaudel B, Bonnetain F, Tijeras-Raballand A, Scriva A, Hickish T, Tabernero J, Van Laethem JL, Banzi M, Maartense E, Shmueli E, Carlsson GU, Scheithauer W, Papamichael D, Moehler M, Landolfi S, Demetter P, Colote S, Tournigand C, Louvet C, Duval A, Flejou JF, de Gramont A. Adjuvant Fluorouracil, Leucovorin, and Oxaliplatin in Stage II to III Colon Cancer: Updated 10-Year Survival and Outcomes According to BRAF Mutation and Mismatch Repair Status of the MOSAIC Study. J Clin Oncol. 2015 Dec 10;33(35):4176-87. doi: 10.1200/JCO.2015.63.4238. Epub 2015 Nov 2. PMID 26527776
- [Background] Andre T, Boni C, Mounedji-Boudiaf L, Navarro M, Tabernero J, Hickish T, Topham C, Zaninelli M, Clingan P, Bridgewater J, Tabah-Fisch I, de Gramont A; Multicenter International Study of Oxaliplatin/5-Fluorouracil/Leucovorin in the Adjuvant Treatment of Colon Cancer (MOSAIC) Investigators. Oxaliplatin, fluorouracil, and leucovorin as adjuvant treatment for colon cancer. N Engl J Med. 2004 Jun 3;350(23):2343-51. doi: 10.1056/NEJMoa032709. PMID 15175436
- [Background] Andre T, Boni C, Navarro M, Tabernero J, Hickish T, Topham C, Bonetti A, Clingan P, Bridgewater J, Rivera F, de Gramont A. Improved overall survival with oxaliplatin, fluorouracil, and leucovorin as adjuvant treatment in stage II or III colon cancer in the MOSAIC trial. J Clin Oncol. 2009 Jul 1;27(19):3109-16. doi: 10.1200/JCO.2008.20.6771. Epub 2009 May 18. PMID 19451431
- [Background] Yothers G, O'Connell MJ, Allegra CJ, Kuebler JP, Colangelo LH, Petrelli NJ, Wolmark N. Oxaliplatin as adjuvant therapy for colon cancer: updated results of NSABP C-07 trial, including survival and subset analyses. J Clin Oncol. 2011 Oct 1;29(28):3768-74. doi: 10.1200/JCO.2011.36.4539. Epub 2011 Aug 22. PMID 21859995
- [Background] Kuebler JP, Wieand HS, O'Connell MJ, Smith RE, Colangelo LH, Yothers G, Petrelli NJ, Findlay MP, Seay TE, Atkins JN, Zapas JL, Goodwin JW, Fehrenbacher L, Ramanathan RK, Conley BA, Flynn PJ, Soori G, Colman LK, Levine EA, Lanier KS, Wolmark N. Oxaliplatin combined with weekly bolus fluorouracil and leucovorin as surgical adjuvant chemotherapy for stage II and III colon cancer: results from NSABP C-07. J Clin Oncol. 2007 Jun 1;25(16):2198-204. doi: 10.1200/JCO.2006.08.2974. Epub 2007 Apr 30. PMID 17470851
- [Background] Schmoll HJ, Tabernero J, Maroun J, de Braud F, Price T, Van Cutsem E, Hill M, Hoersch S, Rittweger K, Haller DG. Capecitabine Plus Oxaliplatin Compared With Fluorouracil/Folinic Acid As Adjuvant Therapy for Stage III Colon Cancer: Final Results of the NO16968 Randomized Controlled Phase III Trial. J Clin Oncol. 2015 Nov 10;33(32):3733-40. doi: 10.1200/JCO.2015.60.9107. Epub 2015 Aug 31. PMID 26324362
- [Background] Haller DG, Tabernero J, Maroun J, de Braud F, Price T, Van Cutsem E, Hill M, Gilberg F, Rittweger K, Schmoll HJ. Capecitabine plus oxaliplatin compared with fluorouracil and folinic acid as adjuvant therapy for stage III colon cancer. J Clin Oncol. 2011 Apr 10;29(11):1465-71. doi: 10.1200/JCO.2010.33.6297. Epub 2011 Mar 7. PMID 21383294
- [Background] Sobrero A, Lonardi S, Rosati G, Di Bartolomeo M, Ronzoni M, Pella N, Scartozzi M, Banzi M, Zampino MG, Pasini F, Marchetti P, Cantore M, Zaniboni A, Rimassa L, Ciuffreda L, Ferrari D, Zagonel V, Maiello E, Barni S, Rulli E, Labianca R; TOSCA Investigators. FOLFOX or CAPOX in Stage II to III Colon Cancer: Efficacy Results of the Italian Three or Six Colon Adjuvant Trial. J Clin Oncol. 2018 May 20;36(15):1478-1485. doi: 10.1200/JCO.2017.76.2187. Epub 2018 Apr 5. PMID 29620994
- [Background] Iveson TJ, Kerr RS, Saunders MP, Cassidy J, Hollander NH, Tabernero J, Haydon A, Glimelius B, Harkin A, Allan K, McQueen J, Scudder C, Boyd KA, Briggs A, Waterston A, Medley L, Wilson C, Ellis R, Essapen S, Dhadda AS, Harrison M, Falk S, Raouf S, Rees C, Olesen RK, Propper D, Bridgewater J, Azzabi A, Farrugia D, Webb A, Cunningham D, Hickish T, Weaver A, Gollins S, Wasan HS, Paul J. 3 versus 6 months of adjuvant oxaliplatin-fluoropyrimidine combination therapy for colorectal cancer (SCOT): an international, randomised, phase 3, non-inferiority trial. Lancet Oncol. 2018 Apr;19(4):562-578. doi: 10.1016/S1470-2045(18)30093-7. PMID 29611518
- [Background] Andre T, Vernerey D, Mineur L, Bennouna J, Desrame J, Faroux R, Fratte S, Hug de Larauze M, Paget-Bailly S, Chibaudel B, Bez J, Dauba J, Louvet C, Lepere C, Dupuis O, Becouarn Y, Mabro M, Egreteau J, Bouche O, Deplanque G, Ychou M, Galais MP, Ghiringhelli F, Dourthe LM, Bachet JB, Khalil A, Bonnetain F, de Gramont A, Taieb J; for PRODIGE investigators, GERCOR, Federation Francaise de Cancerologie Digestive, and UNICANCER. Three Versus 6 Months of Oxaliplatin-Based Adjuvant Chemotherapy for Patients With Stage III Colon Cancer: Disease-Free Survival Results From a Randomized, Open-Label, International Duration Evaluation of Adjuvant (IDEA) France, Phase III Trial. J Clin Oncol. 2018 May 20;36(15):1469-1477. doi: 10.1200/JCO.2017.76.0355. Epub 2018 Apr 5. PMID 29620995
- [Background] Meyerhardt JA, Shi Q, Fuchs CS, Meyer J, Niedzwiecki D, Zemla T, Kumthekar P, Guthrie KA, Couture F, Kuebler P, Bendell JC, Kumar P, Lewis D, Tan B, Bertagnolli M, Grothey A, Hochster HS, Goldberg RM, Venook A, Blanke C, O'Reilly EM, Shields AF. Effect of Celecoxib vs Placebo Added to Standard Adjuvant Therapy on Disease-Free Survival Among Patients With Stage III Colon Cancer: The CALGB/SWOG 80702 (Alliance) Randomized Clinical Trial. JAMA. 2021 Apr 6;325(13):1277-1286. doi: 10.1001/jama.2021.2454. PMID 33821899
- [Background] Souglakos J, Boukovinas I, Kakolyris S, Xynogalos S, Ziras N, Athanasiadis A, Androulakis N, Christopoulou A, Vaslamatzis M, Ardavanis A, Emmanouilides C, Bompolaki I, Kourousis C, Makrantonakis P, Christofyllakis C, Athanasiadis E, Kentepozidis N, Karampeazis A, Katopodi U, Anagnosopoulos A, Papadopoulos G, Prinarakis E, Kalisperi A, Mavroudis D, Georgoulias V. Three- versus six-month adjuvant FOLFOX or CAPOX for high-risk stage II and stage III colon cancer patients: the efficacy results of Hellenic Oncology Research Group (HORG) participation to the International Duration Evaluation of Adjuvant Chemotherapy (IDEA) project. Ann Oncol. 2019 Aug 1;30(8):1304-1310. doi: 10.1093/annonc/mdz193. PMID 31228203
- [Background] Yoshino T, Yamanaka T, Oki E, Kotaka M, Manaka D, Eto T, Hasegawa J, Takagane A, Nakamura M, Kato T, Munemoto Y, Takeuchi S, Bando H, Taniguchi H, Gamoh M, Shiozawa M, Mizushima T, Saji S, Maehara Y, Ohtsu A, Mori M. Efficacy and Long-term Peripheral Sensory Neuropathy of 3 vs 6 Months of Oxaliplatin-Based Adjuvant Chemotherapy for Colon Cancer: The ACHIEVE Phase 3 Randomized Clinical Trial. JAMA Oncol. 2019 Nov 1;5(11):1574-1581. doi: 10.1001/jamaoncol.2019.2572. PMID 31513248
- [Background] Grothey A, Sobrero AF, Shields AF, Yoshino T, Paul J, Taieb J, Souglakos J, Shi Q, Kerr R, Labianca R, Meyerhardt JA, Vernerey D, Yamanaka T, Boukovinas I, Meyers JP, Renfro LA, Niedzwiecki D, Watanabe T, Torri V, Saunders M, Sargent DJ, Andre T, Iveson T. Duration of Adjuvant Chemotherapy for Stage III Colon Cancer. N Engl J Med. 2018 Mar 29;378(13):1177-1188. doi: 10.1056/NEJMoa1713709. PMID 29590544
- [Background] Petrelli F, Labianca R, Zaniboni A, Lonardi S, Galli F, Rulli E, Rosati G, Corallo S, Ronzoni M, Cardellino GG, Mattioli R, Mambrini A, Ciuffreda L, Banzi M, Pusceddu V, Maiello E, Zampino M, Zagonel V, Marchetti P, Corsi D, Rimassa L, Cinieri S, Sobrero A. Assessment of Duration and Effects of 3 vs 6 Months of Adjuvant Chemotherapy in High-Risk Stage II Colorectal Cancer: A Subgroup Analysis of the TOSCA Randomized Clinical Trial. JAMA Oncol. 2020 Apr 1;6(4):547-551. doi: 10.1001/jamaoncol.2019.6486. PMID 32053133
- [Background] Luskin MR, Murakami MA, Manalis SR, Weinstock DM. Targeting minimal residual disease: a path to cure? Nat Rev Cancer. 2018 Apr;18(4):255-263. doi: 10.1038/nrc.2017.125. Epub 2018 Jan 29. PMID 29376520
- [Background] Dasari A, Morris VK, Allegra CJ, Atreya C, Benson AB 3rd, Boland P, Chung K, Copur MS, Corcoran RB, Deming DA, Dwyer A, Diehn M, Eng C, George TJ, Gollub MJ, Goodwin RA, Hamilton SR, Hechtman JF, Hochster H, Hong TS, Innocenti F, Iqbal A, Jacobs SA, Kennecke HF, Lee JJ, Lieu CH, Lenz HJ, Lindwasser OW, Montagut C, Odisio B, Ou FS, Porter L, Raghav K, Schrag D, Scott AJ, Shi Q, Strickler JH, Venook A, Yaeger R, Yothers G, You YN, Zell JA, Kopetz S. ctDNA applications and integration in colorectal cancer: an NCI Colon and Rectal-Anal Task Forces whitepaper. Nat Rev Clin Oncol. 2020 Dec;17(12):757-770. doi: 10.1038/s41571-020-0392-0. Epub 2020 Jul 6. PMID 32632268
- [Background] Tie J, Wang Y, Tomasetti C, Li L, Springer S, Kinde I, Silliman N, Tacey M, Wong HL, Christie M, Kosmider S, Skinner I, Wong R, Steel M, Tran B, Desai J, Jones I, Haydon A, Hayes T, Price TJ, Strausberg RL, Diaz LA Jr, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating tumor DNA analysis detects minimal residual disease and predicts recurrence in patients with stage II colon cancer. Sci Transl Med. 2016 Jul 6;8(346):346ra92. doi: 10.1126/scitranslmed.aaf6219. PMID 27384348
- [Background] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Background] Tie J, Cohen JD, Wang Y, Christie M, Simons K, Lee M, Wong R, Kosmider S, Ananda S, McKendrick J, Lee B, Cho JH, Faragher I, Jones IT, Ptak J, Schaeffer MJ, Silliman N, Dobbyn L, Li L, Tomasetti C, Papadopoulos N, Kinzler KW, Vogelstein B, Gibbs P. Circulating Tumor DNA Analyses as Markers of Recurrence Risk and Benefit of Adjuvant Therapy for Stage III Colon Cancer. JAMA Oncol. 2019 Dec 1;5(12):1710-1717. doi: 10.1001/jamaoncol.2019.3616. PMID 31621801
- [Background] Barault L, Amatu A, Siravegna G, Ponzetti A, Moran S, Cassingena A, Mussolin B, Falcomata C, Binder AM, Cristiano C, Oddo D, Guarrera S, Cancelliere C, Bustreo S, Bencardino K, Maden S, Vanzati A, Zavattari P, Matullo G, Truini M, Grady WM, Racca P, Michels KB, Siena S, Esteller M, Bardelli A, Sartore-Bianchi A, Di Nicolantonio F. Discovery of methylated circulating DNA biomarkers for comprehensive non-invasive monitoring of treatment response in metastatic colorectal cancer. Gut. 2018 Nov;67(11):1995-2005. doi: 10.1136/gutjnl-2016-313372. Epub 2017 Oct 5. PMID 28982739
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Middleton MR, Grob JJ, Aaronson N, Fierlbeck G, Tilgen W, Seiter S, Gore M, Aamdal S, Cebon J, Coates A, Dreno B, Henz M, Schadendorf D, Kapp A, Weiss J, Fraass U, Statkevich P, Muller M, Thatcher N. Randomized phase III study of temozolomide versus dacarbazine in the treatment of patients with advanced metastatic malignant melanoma. J Clin Oncol. 2000 Jan;18(1):158-66. doi: 10.1200/JCO.2000.18.1.158. PMID 10623706
- [Background] Fu D, Calvo JA, Samson LD. Balancing repair and tolerance of DNA damage caused by alkylating agents. Nat Rev Cancer. 2012 Jan 12;12(2):104-20. doi: 10.1038/nrc3185. PMID 22237395
- [Background] Amatu A, Sartore-Bianchi A, Moutinho C, Belotti A, Bencardino K, Chirico G, Cassingena A, Rusconi F, Esposito A, Nichelatti M, Esteller M, Siena S. Promoter CpG island hypermethylation of the DNA repair enzyme MGMT predicts clinical response to dacarbazine in a phase II study for metastatic colorectal cancer. Clin Cancer Res. 2013 Apr 15;19(8):2265-72. doi: 10.1158/1078-0432.CCR-12-3518. Epub 2013 Feb 19. PMID 23422094
- [Background] Hochhauser D, Glynne-Jones R, Potter V, Gravalos C, Doyle TJ, Pathiraja K, Zhang Q, Zhang L, Sausville EA. A phase II study of temozolomide in patients with advanced aerodigestive tract and colorectal cancers and methylation of the O6-methylguanine-DNA methyltransferase promoter. Mol Cancer Ther. 2013 May;12(5):809-18. doi: 10.1158/1535-7163.MCT-12-0710. Epub 2013 Feb 26. PMID 23443801
- [Background] Pietrantonio F, Perrone F, de Braud F, Castano A, Maggi C, Bossi I, Gevorgyan A, Biondani P, Pacifici M, Busico A, Gariboldi M, Festinese F, Tamborini E, Di Bartolomeo M. Activity of temozolomide in patients with advanced chemorefractory colorectal cancer and MGMT promoter methylation. Ann Oncol. 2014 Feb;25(2):404-8. doi: 10.1093/annonc/mdt547. Epub 2013 Dec 29. PMID 24379162
- [Background] Pietrantonio F, de Braud F, Milione M, Maggi C, Iacovelli R, Dotti KF, Perrone F, Tamborini E, Caporale M, Berenato R, Leone G, Pellegrinelli A, Bossi I, Festinese F, Federici S, Di Bartolomeo M. Dose-Dense Temozolomide in Patients with MGMT-Silenced Chemorefractory Colorectal Cancer. Target Oncol. 2016 Jun;11(3):337-43. doi: 10.1007/s11523-015-0397-2. PMID 26538496
- [Background] Amatu A, Barault L, Moutinho C, Cassingena A, Bencardino K, Ghezzi S, Palmeri L, Bonazzina E, Tosi F, Ricotta R, Cipani T, Crivori P, Gatto R, Chirico G, Marrapese G, Truini M, Bardelli A, Esteller M, Di Nicolantonio F, Sartore-Bianchi A, Siena S. Tumor MGMT promoter hypermethylation changes over time limit temozolomide efficacy in a phase II trial for metastatic colorectal cancer. Ann Oncol. 2016 Jun;27(6):1062-1067. doi: 10.1093/annonc/mdw071. Epub 2016 Feb 24. PMID 26916096
- [Background] Calegari MA, Inno A, Monterisi S, Orlandi A, Santini D, Basso M, Cassano A, Martini M, Cenci T, de Pascalis I, Camarda F, Barbaro B, Larocca LM, Gori S, Tonini G, Barone C. A phase 2 study of temozolomide in pretreated metastatic colorectal cancer with MGMT promoter methylation. Br J Cancer. 2017 May 9;116(10):1279-1286. doi: 10.1038/bjc.2017.109. Epub 2017 Apr 20. PMID 28427088
- [Background] Morano F, Corallo S, Niger M, Barault L, Milione M, Berenato R, Moretto R, Randon G, Antista M, Belfiore A, Raimondi A, Nichetti F, Martinetti A, Battaglia L, Perrone F, Pruneri G, Falcone A, Di Bartolomeo M, de Braud F, Di Nicolantonio F, Cremolini C, Pietrantonio F. Temozolomide and irinotecan (TEMIRI regimen) as salvage treatment of irinotecan-sensitive advanced colorectal cancer patients bearing MGMT methylation. Ann Oncol. 2018 Aug 1;29(8):1800-1806. doi: 10.1093/annonc/mdy197. PMID 29860358
- [Background] Pietrantonio F, Lobefaro R, Antista M, Lonardi S, Raimondi A, Morano F, Mosconi S, Rimassa L, Murgioni S, Sartore-Bianchi A, Tomasello G, Longarini R, Farina G, Petrelli F, Gori S, Randon G, Corallo S, Pagani F, Guarini V, Palermo F, Martinetti A, Macagno M, Barault L, Perrone F, Tamborini E, Milione M, Di Nicolantonio F, Di Maio M, Fuca G, Di Bartolomeo M, de Braud F. Capecitabine and Temozolomide versus FOLFIRI in RAS-Mutated, MGMT-Methylated Metastatic Colorectal Cancer. Clin Cancer Res. 2020 Mar 1;26(5):1017-1024. doi: 10.1158/1078-0432.CCR-19-3024. Epub 2019 Nov 18. PMID 31740551
- [Background] Houghton PJ, Stewart CF, Cheshire PJ, Richmond LB, Kirstein MN, Poquette CA, Tan M, Friedman HS, Brent TP. Antitumor activity of temozolomide combined with irinotecan is partly independent of O6-methylguanine-DNA methyltransferase and mismatch repair phenotypes in xenograft models. Clin Cancer Res. 2000 Oct;6(10):4110-8. PMID 11051264
- [Background] Pourquier P, Waltman JL, Urasaki Y, Loktionova NA, Pegg AE, Nitiss JL, Pommier Y. Topoisomerase I-mediated cytotoxicity of N-methyl-N'-nitro-N-nitrosoguanidine: trapping of topoisomerase I by the O6-methylguanine. Cancer Res. 2001 Jan 1;61(1):53-8. PMID 11196197
- [Background] Pommier Y. Topoisomerase I inhibitors: camptothecins and beyond. Nat Rev Cancer. 2006 Oct;6(10):789-802. doi: 10.1038/nrc1977. PMID 16990856
- [Background] Sartore-Bianchi A, Pietrantonio F, Amatu A, Milione M, Cassingena A, Ghezzi S, Caporale M, Berenato R, Falcomata C, Pellegrinelli A, Bardelli A, Nichelatti M, Tosi F, De Braud F, Di Nicolantonio F, Barault L, Siena S. Digital PCR assessment of MGMT promoter methylation coupled with reduced protein expression optimises prediction of response to alkylating agents in metastatic colorectal cancer patients. Eur J Cancer. 2017 Jan;71:43-50. doi: 10.1016/j.ejca.2016.10.032. Epub 2016 Dec 18. PMID 27997874
- [Background] Schwartz S, Szeto C, Tian Y, Cecchi F, Corallo S, Calegari MA, Di Bartolomeo M, Morano F, Raimondi A, Fuca G, Martinetti A, De Pascalis I, Martini M, Belfiore A, Milione M, Orlandi A, Barault L, Barone C, de Braud F, Di Nicolantonio F, Benz S, Hembrough T, Pietrantonio F. Refining the selection of patients with metastatic colorectal cancer for treatment with temozolomide using proteomic analysis of O6-methylguanine-DNA-methyltransferase. Eur J Cancer. 2019 Jan;107:164-174. doi: 10.1016/j.ejca.2018.11.016. Epub 2018 Dec 19. PMID 30579113
- [Background] Pietrantonio F, Randon G, Romagnoli D, Di Donato S, Benelli M, de Braud F. Biomarker-guided implementation of the old drug temozolomide as a novel treatment option for patients with metastatic colorectal cancer. Cancer Treat Rev. 2020 Jan;82:101935. doi: 10.1016/j.ctrv.2019.101935. Epub 2019 Nov 28. PMID 31821983
- [Background] Germano G, Lamba S, Rospo G, Barault L, Magri A, Maione F, Russo M, Crisafulli G, Bartolini A, Lerda G, Siravegna G, Mussolin B, Frapolli R, Montone M, Morano F, de Braud F, Amirouchene-Angelozzi N, Marsoni S, D'Incalci M, Orlandi A, Giraudo E, Sartore-Bianchi A, Siena S, Pietrantonio F, Di Nicolantonio F, Bardelli A. Inactivation of DNA repair triggers neoantigen generation and impairs tumour growth. Nature. 2017 Dec 7;552(7683):116-120. doi: 10.1038/nature24673. Epub 2017 Nov 29. PMID 29186113
- [Background] Morano F, Corallo S, Lonardi S, Raimondi A, Cremolini C, Rimassa L, Murialdo R, Zaniboni A, Sartore-Bianchi A, Tomasello G, Racca P, Clavarezza M, Adamo V, Perrone F, Gloghini A, Tamborini E, Busico A, Martinetti A, Palermo F, Loupakis F, Milione M, Fuca G, Di Bartolomeo M, de Braud F, Pietrantonio F. Negative Hyperselection of Patients With RAS and BRAF Wild-Type Metastatic Colorectal Cancer Who Received Panitumumab-Based Maintenance Therapy. J Clin Oncol. 2019 Nov 20;37(33):3099-3110. doi: 10.1200/JCO.19.01254. Epub 2019 Sep 20. PMID 31539295
- [Background] Siravegna G, Mussolin B, Buscarino M, Corti G, Cassingena A, Crisafulli G, Ponzetti A, Cremolini C, Amatu A, Lauricella C, Lamba S, Hobor S, Avallone A, Valtorta E, Rospo G, Medico E, Motta V, Antoniotti C, Tatangelo F, Bellosillo B, Veronese S, Budillon A, Montagut C, Racca P, Marsoni S, Falcone A, Corcoran RB, Di Nicolantonio F, Loupakis F, Siena S, Sartore-Bianchi A, Bardelli A. Clonal evolution and resistance to EGFR blockade in the blood of colorectal cancer patients. Nat Med. 2015 Jul;21(7):827. doi: 10.1038/nm0715-827b. No abstract available. PMID 26151329
- [Background] Arena S, Siravegna G, Mussolin B, Kearns JD, Wolf BB, Misale S, Lazzari L, Bertotti A, Trusolino L, Adjei AA, Montagut C, Di Nicolantonio F, Nering R, Bardelli A. MM-151 overcomes acquired resistance to cetuximab and panitumumab in colorectal cancers harboring EGFR extracellular domain mutations. Sci Transl Med. 2016 Feb 3;8(324):324ra14. doi: 10.1126/scitranslmed.aad5640. PMID 26843189